CLINICAL TRIAL: NCT00274898
Title: Phase II Randomized Study Evaluting the Effect of Celecoxib as Maintenance Treatment of Stage IIIb Non-Small Cell Lung Cancer That Reponded or is Stable After Radiochemotherapy
Brief Title: Celecoxib or Observation After Radiation Therapy and Chemotherapy in Treating Patients With Stage II or Stage III Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454352; GERCOR-B03-1; EU-20572; SANOFI-GERCOR-B03-1; PFIZER-GERCOR-B03-1
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-09

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Docetaxel; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: celecoxib
Drug: docetaxel
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving celecoxib after radiation therapy and chemotherapy may kill any tumor cells that remain after radiation therapy and chemotherapy. Sometimes, after radiation therapy and chemotherapy, the tumor may not need additional treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This randomized phase II trial is studying celecoxib to see how well it works compared to observation in treating patients who have undergone radiation therapy and chemotherapy for stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the time to progression in patients with stage II-IIIB non-small cell lung cancer treated with celecoxib vs observation after treatment with chemoradiotherapy.

Secondary

* Compare the 2-year survival rate of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare weight changes and objective response in patients treated with these regimens.
* Compare tolerability of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, ECOG performance status (0-1 vs 2), and total dose of radiotherapy (65 Gy vs 60 Gy).

All patients undergo radiotherapy 5 days a week for 7.5 weeks. Patients also receive docetaxel IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Three weeks after the completion of radiotherapy, patients receive docetaxel alone IV over 30 minutes on days 1 and 22. Three weeks later, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are observed every 3 months for 1 year and then every 6 months for 1 year.
* Arm II: Patients receive oral celecoxib twice daily for up to 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 3 months for 1 year, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer meeting ≥ 1 of the following criteria:

  * Stage IIIB disease
  * Stage II or IIIA disease, meeting the following criteria:

    * Considered nonresectable
    * Pleural effusion present
* Measurable disease
* Must have received a prior regimen of radiotherapy and chemotherapy comprising docetaxel and carboplatin
* Tumor volume must be able to be encompassed in the radiation field

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 12 weeks
* Cardiac function compatible with radiotherapy
* Neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.25 times ULN
* AST and ALT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* No other malignancy in the past 10 years except basal cell skin cancer or carcinoma in situ of the cervix
* No active infection
* No inflammatory bowel disease
* No severe congestive heart failure
* No severe hepatic disease defined as albumin < 25 g/L or Child-Pugh score ≥ 10
* No severe renal disease defined as creatinine clearance < 30 mL/min
* No known hypersensitivity to sulfonamides, the study or it's excipients, or polysorbate 80
* No known hypersensitivity of NSAIDs, salicylic acid, or cyclo-oxygenase-2 inhibitors
* No familial, social, geographical, or psychological condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since participation in another clinical study
* More than 1 month since prior therapy for gastrointestinal ulcers
* No concurrent fluconazole, ketoconazole, lithium, or dextromethorphan
* No other concurrent anticancer treatment including chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or biologic response modifier therapy
* No concurrent aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)

  * Low-dose aspirin or NSAIDs for a duration of ≤ 1 week during the past 3 months allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-05

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
2-year survival rate
Quality of life
Weight changes
Objective response
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jean F. Morere, MD, Study Chair — Hopital Avicenne
Locations (15):
- France (15):
  - Hopital Avicenne, Bobigny
  - Centre Medical de Forcilles Hopital Prive, Ferroles Attilly
  - Clinique du Petit Colmouilins, Harfleur
  - Clinique Victor Hugo, Le Mans
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - American Hospital of Paris, Neuilly-sur-Seine
  - Clinique De Valdegour, Nîmes
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - Clinique les Bleuets, Reims
  - Polyclinique De Courlancy, Reims
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Hospitalier Sud-Reiunion, Saint-Pierre
  - Clinique Sainte Clotilde, Sainte Clotilde